CLINICAL TRIAL: NCT05749224
Title: Turkish Validity and Reliability of The Helkimo Index for Diagnosis of Temporomandibular Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: DenizOzluer
Record Dates: First submitted 2022-12-24; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-12

CONDITIONS: Temporomandibular Disorder
Keywords: helkimo index; temporomandibular disorders; Turkish validity and reliability
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Who Have Temporomandibular Joint Disorder (Experimental): Helkimo index will be applied to the patients have temporomandibular disorder.
  Interventions: Diagnostic Test: Helkimo Index
- Healthy Controls (Experimental): Helkimo index will be applied to healthy people.
  Interventions: Diagnostic Test: Helkimo Index

INTERVENTIONS:
Diagnostic Test: Helkimo Index — Helkimo Index is comprised of five items, with each assessment having three possible answers, scored as 0, 1 or 5. The first item is related to the limitation in the range of jaw movement. The second item evaluates the alterations of joint function that produce deviations, sounds and/or joint locks or blockages; the third item evaluates the presence of pain when performing some movements; the fourth item evaluates muscular pain in the masticatory muscles; and the fifth item evaluates the presence of discomfort or pain in the prearticular area of the temporomandibular joint (TMJ) through palpation. From the sum of the 5 items, we identify no TMJ involvement if the score is 0, mild TMJ involvement when the score ranges from 1 to 9, moderate TMJ involvement if the score ranges between 10 and 19 and severe TMJ involvement for a score between 20 and 25.

SUMMARY:
Helkimo Index evaluates movement, joint function, pain and musculature, providing a quick general overview that could be very useful at different levels of care. The aim of this study is to investigate the validity and reliability of the Turkish version of the Helkimo index. Registration of subjective symptoms applying for the Helkimo Index required a questionnaire-based survey. Questionnaire comprised two parts: Anamnestic component which includes answers to questions in "yes" or "no". Clinical dysfunction part comprised clinical examination. Method: Turkish translation of Helkimo index will be made. The sample will consist of 100 subjects, 50 TMD patients and 50 healthy controls. the patients will be selected, demographic data were recorded: age, sex, height, weight, body mass index (BMI), educational level, work situation, smoking status, alcoholic habits and physical activity. Helkimo Index is comprised of five items, with each assessment having three possible answers, scored as 0, 1 or 5. The first item is related to the limitation in the range of jaw movement. The second item evaluates the alterations of joint function that produce deviations, sounds and/or joint locks or blockages; the third item evaluates the presence of pain when performing some movements; the fourth item evaluates muscular pain in the masticatory muscles; and the fifth item evaluates the presence of discomfort or pain in the prearticular area of the temporomandibular joint (TMJ) through palpation. From the sum of the 5 items, we identify no TMJ involvement if the score is 0, mild TMJ involvement when the score ranges from 1 to 9, moderate TMJ involvement if the score ranges between 10 and 19 and severe TMJ involvement for a score between 20 and 25. The Numerical Pain-Rating Scale (NPRS) test, disability, the Neck Disability Index test, the Dizziness Handicap Inventory (DHI), the Headache Impact Test (HIT-6) and 12-item Short-Form Health Survey (SF-12) will be assessed. Correlation will be made between the Helkimo index and these rating scales.

DETAILED DESCRIPTION:
Temporomandibular disorder (TMD) is a wide-ranging term used to describe a number of related disorders involving the temporomandibular joint (TMJ), masticatory muscles, and occlusion, with common symptoms such as pain, restricted movement, muscle tenderness, and intermittent joint sounds. TMDs can also be defined as a collective term for conditions that involve pain and/or dysfunction of the TMJ and the related structures. The Helkimo Clinical Dysfunction Index (HCDI) has been widely used for the clinical diagnosis of TMDs. It is a simple and quick test that assesses limitations of mandibular movement, pain and joint function. However, the studies that analyze the reliability and validity of this tool are old, used a very small sample, applied incorrect statistical techniques and were limited to the analysis of a single clinometric property. The diagnostic validity of the HCDI was measured according to diagnostic criteria for temporomandibular disorders (DC/TMDs) protocol, which is the gold-standard diagnostic test for TMD. The DC/TMD protocol is composed of 12 items that assess muscle and joint pain, pain during jaw movement, headache, bites, noise, obstacles or blockages during jaw movement and discomfort in the palpation of the muscles of the temporomandibular joint. Finally, a diagnostic tree is used to specify a diagnostic result. The DC/TMD protocol has a sensitivity of 86%, a specificity of 98% and an inter-examination reliability of 85%. The main measure was the HCDI. The instrument is comprised of five items, with each assessment having three possible answers, scored as 0, 1 or 5. The first item is related to the limitation in the range of jaw movement. The second item evaluates the alterations of joint function that produce deviations, sounds and/or joint locks or blockages; the third item evaluates the presence of pain when performing some movements; the fourth item evaluates muscular pain in the masticatory muscles; and the fifth item evaluates the presence of discomfort or pain in the prearticular area of the temporomandibular joint (TMJ) through palpation. From the sum of the 5 items, we identify no TMJ involvement if the score is 0, mild TMJ involvement when the score ranges from 1 to 9, moderate TMJ involvement if the score ranges between 10 and 19 and severe TMJ involvement for a score between 20 and 25.

Pain perception will be evaluated by the Numerical Pain-Rating Scale (NPRS) test. The subjects indicate their perceived pain with a number between 0 (no pain) and 10 (the worst pain possible). This tool is used to quantify both the neck and the temporomandibular joint and is the pain assessment.

To evaluate the possibility of associate neck disability, the Neck Disability Index test will be used; it is a 10-question survey, with answers being reported as a number between 0 and 5. For each question, a score of 0 refers to the total absence of disability, while a score of 5 refers to total disability. In this line, a total score between 0 and 5 indicates absence of disability, 5-14 points indicate low disability, 15-24 point indicates moderate disability and 35-50 points indicate great disability.

The presence of vertigo and balance problems will be assessed by the Dizziness Handicap Inventory (DHI). This questionnaire is composed of 25 questions that can be answered with yes, no or sometimes, scoring 4, 0 and 2 points, respectively. This questionnaire assesses physical, emotional and functional dimensions, each of which has an independent score in addition to the total score.

Headache-associated symptoms will be measured with the Headache Impact Test (HIT-6), which is an evaluation questionnaire consisting of six questions that can be answered with usual, almost always, sometimes, rarely and never, with a total score between 36 and 78 points.

Finally, the quality of life will be assessed using the 12-item Short-Form Health Survey (SF-12). This questionnaire is the short version of the SF-36 and retains its self-administered form. It results in a Mental Component Summary score and a Physical Component Summary score (PCS-12), differentiating between the two components of the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18

Exclusion Criteria:

* History of TMJ surgery, having neuromuscular disorders, having vestibular symptoms which affects balance

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-26 (Estimated)

PRIMARY OUTCOMES:
Helkimo Index for Diagnosis of Temporomandibular Disorders | 3 months
  Turkish Validity and Reliability Study
Questionnaire for Anamnestic Component of Helkimo Index | 3 months
  It is an anamnestic component questionnaire consisting of 8 different questions asked verbally to the participants and forming the first part of the Helkimo index.
Clinical Dysfunction Component of Helkimo Index | 3 months
  It is a clinical dysfunction questionnaire that constitutes the second part of the helkimo index, in which the temporamandibular joint of the participants is evaluated physically with 5 different parameters.

SECONDARY OUTCOMES:
SF-12 | 3 months
  Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Elif Tugce Cil, PhD, Study Director — Yeditepe University

IPD SHARING:
Plan to Share IPD: Yes
Cultural adaptation of the Helkimo index to Turkish society will be done.
Supporting Information: Study Protocol, CSR
Time Frame: In 2023 - Infinite Access
Access Criteria: No access criteria

REFERENCES:
- See also: Validity and Reliability of the Helkimo Clinical Dysfunction Index for the Diagnosis of Temporomandibular Disorders — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8000811/pdf/diagnostics-11-00472.pdf
- See also: Analysis of Helkimo index for temporomandibular disorder diagnosis in the dental students of Faridabad city: A cross-sectional study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5308067/pdf/JIPS-17-48.pdf